CLINICAL TRIAL: NCT06054334
Title: Relevance of Isoniazid Dosage in Adults Treated for Tuberculosis
Acronym: ISOBK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2023_843_0003
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Tuberculosis
Keywords: Isoniazid; tuberculosis; acetylation
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tuberculosis is the third leading infectious killer. In 2021, an estimated 10,6 million people fell ill with tuberculosis worldwide. Drug resistance emerges with the increase of antibiotherapy use. Among the four antimicrobial drugs used for tuberculosis, isoniazid is a first line treatment. It has a bactericidal activity against the tuberculosis complex. Nevertheless, the hepatic metabolism of isoniazid shows variation between individuals. There is a real risk of hepatotoxicity and neurotoxicity induced by isoniazid. The peak measurement (Cmax) of serum isoniazid is recommended to adjust the treatment and to allow recovery. Moreover, several samples allow a kinetics of isoniazid elimination so as to distinguish slow and fast acetylators. Few data are available on isoniazid acetylation. It could be useful to know the proportion of patients treated by isoniazid at a standard dose, associated with a risk of overdosing or underdosing. Inadequate exposures should be studied to understand if there is an impact in the medical care.

ELIGIBILITY:
Inclusion Criteria:

* to be an adult,
* to have a diagnosis of tuberculosis

Exclusion Criteria:

* pregnancy,
* disagreement to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical study aims to examine the relevance of isoniazid dosage in adults treated for tuberculosis.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Serum isoniazid Cmax | between day 15 and day 30
  : Serum isoniazid Cmax in the standards, (i.e., between 3 et 6 µg/ml measured at 1h or 2h).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No